CLINICAL TRIAL: NCT03043339
Title: Characterization Of the Intestinal Microbiome Evolution After Kidney Transplant Donation or Receipt
Acronym: COMET-DR
Status: Terminated | Type: Observational
Why Stopped: Study halted prematurely due to lack of funding.
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen S. Kraft, Associate Professor, Emory University
Other Study IDs: IRB00092450; 16IPA1609418 (Other Grant/Funding Number: Centers for Disease Control and Prevention (CDC)); 16IPA1609428 (Other Grant/Funding Number: Centers for Disease Control and Prevention (CDC)); CDC-IRB00092450 (Other: Centers for Disease Control and Prevention (CDC))
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Renal Transplant
Keywords: Microbiota composition; Kidney transplant recipient; Kidney transplant donor; Antibiotics; Drug resistance; Transplantation surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected through anal swabs and stool samples will be stored until DNA extraction can occur. DNA analysis of the microbiome will occur; DNA of the participants will not be examined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Renal transplant recipient: Participants who are scheduled for a planned renal transplant as the recipient of the kidney.
  All participants will complete the following interventions:
  * Stool Specimen Collection
  * Anal Swab Sampling
  * Short Diet Assessment (SDA)
  * NHANES Dietary Screener Questionnaire (DSQ)
  Interventions: Other: Stool Specimen Collection; Other: Anal Swab Sampling; Other: Short Diet Assessment (SDA); Other: NHANES Dietary Screener Questionnaire (DSQ)
- Renal transplant donor: Participants who are scheduled for a planned renal transplant as the donor of the kidney.
  All participants will complete the following interventions:
  * Stool Specimen Collection
  * Anal Swab Sampling
  * Short Diet Assessment (SDA)
  * NHANES Dietary Screener Questionnaire (DSQ)
  Interventions: Other: Stool Specimen Collection; Other: Anal Swab Sampling; Other: Short Diet Assessment (SDA); Other: NHANES Dietary Screener Questionnaire (DSQ)

INTERVENTIONS:
Other: Stool Specimen Collection — Participants will provide a stool sample at baseline (pre-operation) and 30 days after the transplant operation. Stool specimens will be self-collected by the participant.
Other: Anal Swab Sampling — Anal swabs will be collected prior to surgery (baseline) and at post-operation days 2, 15, and 30. Participants whose planned hospitalization duration is extended from the pre-surgical plan will have an additional, optional, anal swab collected 2 days prior to their anticipated hospital discharge date. Anal swabs will be collected by the study team, except for the standard of care post-operative appointment (30 days after the operation) for the living donors who will collect their own samples.
Other: Short Diet Assessment (SDA) — The study coordinator will administer the Short Diet Assessment (SDA) to participants prior to surgery at baseline and post-operation days 2, 15, and 30. Participants whose planned hospital length of stay is extended from the pre-surgical plan will complete the questionnaire 2 days prior to their anticipated hospital discharge date.
Other: NHANES Dietary Screener Questionnaire (DSQ) — The National Health and Nutrition Examination Survey (NHANES) 2009-2010 Dietary Screener Questionnaire will be completed on Post-Operative Day 2. The questionnaire asks about foods consumed during the past 30 days. There are 25 items on the questionnaire and additional questions may be asked depending on responses provided. The questionnaire will be self-administered or administered by a study team member.

SUMMARY:
This is a hypothesis-generating pilot study. The intent is to model the impact of perioperative practices on the intestinal microbiome and possibly associate these conditions with the final microbiome status (e.g., number of resistance genes and diversity associated with perioperative practices and preoperative microbiome status). Participants will include individuals who are having surgery to either receive or donate a kidney. To determine the diversity change of the intestinal microbiota over time, rectal swabs will be collected before surgery and at several time points after surgery, with the last swab collected 30 days after surgery.

This pilot study is to obtain preliminary data to support the rationale and design for a subsequent clinical trial. This study is designed to understand the intestinal microbiota diversity in the setting of renal transplant surgery and the clinical significance of antibiotic use and the associated resistome (collection of all antibiotic resistance genes and precursors within a sample).

DETAILED DESCRIPTION:
The emergence of multidrug resistant organisms (MDROs) is a growing threat to global public health and is associated with high morbidity and mortality in both the general and solid organ transplant population. Intestinal microbiota diversity can provide functional and spatial barriers to bacterial and fungal MDRO colonization, and loss of diversity is associated with increased MDRO colonization. Dysbiosis is a state of loss of microbiota diversity and a single antibiotic treatment course can cause significant disruption in microbiota diversity, even in otherwise healthy individuals. This disruption can promote the growth of pathogenic and multidrug-resistant bacteria and fungi. Transplant patients, in particular, are at increased risk of colonization and infection with MDRO because of immunomodulatory therapies, healthcare exposure, increased antibiotic exposure and surgical manipulation of mucosa. Furthermore, chronic kidney disease and dialysis therapy leading up to transplant has been shown to be associated with alterations in both the intestinal and periodontal microbiome. Understanding the evolution of the disruption in the intestinal microbiome in both kidney transplant recipients and healthy kidney transplant donors during the time of transplant surgical prophylaxis will give valuable insight into further avenues for research and possible interventions that may mitigate the risk of MDRO colonization.

This is a prospective, observational, and non-interventional pilot study which aims to enroll 100 adult renal transplant recipients and 100 adult renal transplant donors. Participants will provide stool samples and anal swab samples, and will complete dietary questionnaires. Participants may also choose to take part in an optional sub-study which involves banking leftover stool for future research use.

The diversity change of the intestinal microbiota over time will be assessed at the screening visit, Post-Operative Day 2; Post-Discharge Day 15 and Post-Discharge Day 30. Participants will be followed by way of medical record review for 24 weeks post-surgery.

This study is designed to understand the intestinal microbiota diversity in the setting of renal transplant surgery and the clinical significance of antibiotic use and the associated resistome (collection of all antibiotic resistance genes and precursors within a sample). Information learned from this study will be used to guide the design of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Ability and willingness to comply with study protocol requirements.
* Completed Verbal Screening Form
* Planned kidney donation or planned receipt of a living donor kidney transplant within 28 days from time of written informed consent.
* If performance status is known, a score of any of the following:

  * American Society of Anesthesia (ASA) classification of I (a normal healthy patient), II (a patient with mild systemic disease) or III (a patient with severe systemic disease)
  * Eastern Cooperative Oncology Group (ECOG) Status Scale grade of 0 (normal activity), 1 (symptoms, but ambulatory) or 2 (in bed <50% of the time)
  * Karnofsky Performance Scale (KPS) of 50% (requires considerable assistance and frequent medical care) to 100% (normal, no complaints, no evidence of disease)
* English speaking.

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, might interfere with study objectives or limit compliance with study requirements, including but not limited to:

  * Known active intravenous drug or alcohol abuse
  * Psychiatric illness
  * Social situation
* Planned or actual receipt of a deceased donor kidney transplant.
* Prior kidney transplant that still requires active immunosuppressive treatment or intervention.
* Presence of diverting ileostomy or colostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients and living donors
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Change in microbiota composition | Baseline to Postoperative Day 30
  To understand the overall impact of surgical prophylaxis on intestinal microbiota composition in the setting of renal transplant surgery, the distribution and relative abundance of bacterial and fungal taxa for each collected sample will be described. A genus of strain will be considered predominant if it represents at least 30% of all genus or strains of microbiota within the stool sample.
Change in microbiota diversity | Baseline to Postoperative Day 30
  To understand the overall impact of surgical prophylaxis on intestinal microbiota diversity in the setting of renal transplant surgery, measures of α- and β-diversity of the intestinal microbiota will be utilized. The maximum percentage of all genes identified included within the same taxon will be determined from each stool sample.
Change in microbiota taxonomy | Baseline to Postoperative Day 30
  To understand the overall impact of surgical prophylaxis on intestinal microbiota taxonomy, in the setting of renal transplant surgery, the collected specimens will be used for taxonomic composition determination of bacteria and fungi. Whole genome shotgun metagenomic sequencing will be performed on an Illumina Miseq (or HiSeq). A short read mapper will be used to screen out and discard human sequences from each stool sample and subsequently Metaphlan and KRAKEN are used for taxonomic composition determination.
Change in microbiota resistome | Baseline to Postoperative Day 30
  To understand the overall impact of surgical prophylaxis on intestinal microbiota resistance, in the setting of renal transplant surgery, the study samples collected will be used to provide a summary of the overall number and diversity of bacterial and fungal resistance genes, including any new acquisition.

SECONDARY OUTCOMES:
Microbiota composition in renal dialysis patients | Baseline
  To understand the intestinal microbiota composition in patients receiving renal dialysis, the distribution and relative abundance of bacterial and fungal taxa for each collected sample will be described. A genus of strain will be considered predominant if it represents at least 30% of all genus or strains of microbiota within the stool sample collected at baseline (prior to renal transplant).
Microbiota diversity in renal dialysis patients | Baseline
  To understand the intestinal microbiota Alpha and Beta diversity in patients receiving renal dialysis, the maximum percentage of all genes identified included within the same taxon will be determined from the study samples collected at baseline (prior to renal transplant).
Microbiota resistome in renal dialysis patients | Baseline
  To understand the intestinal microbiota resistance in patients receiving renal dialysis, the study samples collected at baseline (prior to renal transplant) will be used to provide a summary of the overall number and diversity of bacterial resistance genes.

OTHER OUTCOMES:
Compare microbiota composition of donors and recipients | Baseline
  The exploratory objective of this study is to characterize the similarities and differences in intestinal microbiota between living donor and recipients at the baseline time point. The distribution and relative abundance of bacterial and fungal taxa for each baseline sample (prior to renal transplant) will be described. A genus of strain will be considered predominant if it represents at least 30% of all genus or strains of microbiota within the stool sample.
Compare microbiota diversity of donors and recipients | Baseline
  The exploratory objective of this study is to characterize the similarities and differences in intestinal microbiota between living donor and recipients at the baseline time point. The maximum percentage of all genes identified included within the same taxon will be determined from each stool sample collected prior to renal transplant.
Compare microbiota taxonomy of donors and recipients | Baseline
  The exploratory objective of this study is to characterize the similarities and differences in intestinal microbiota between living donor and recipients at the baseline time point. The study samples collected will be used for taxonomic composition determination of bacteria and fungi. Whole genome shotgun metagenomic sequencing will be performed on an Illumina Miseq (or HiSeq). A short read mapper will be used to screen out and discard human sequences from each stool sample and subsequently Metaphlan and KRAKEN are used for taxonomic composition determination.
Compare microbiota resistome of donors and recipients | Baseline
  The exploratory objective of this study is to characterize the similarities and differences in intestinal microbiota between living donor and recipients at the baseline time point. The study samples collected will be used to provide a summary of the overall number and diversity of bacterial and fungal resistance genes, including any new acquisition.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen S Kraft, MD, MSc, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - The Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT03043339/ICF_000.pdf